CLINICAL TRIAL: NCT05891496
Title: A Randomised Double-blind Placebo-controlled Clinical Study Investigating the Effects of Semaglutide s.c. Once-weekly Versus Placebo on Central and Peripheral Inflammation in Participants With Alzheimer's Disease
Brief Title: A Research Study Looking at the Effect of Semaglutide on the Immune System and Other Biological Processes in People With Alzheimer's Disease
Status: Active, not recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: Novo Nordisk A/S (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: NN6535-7519; U1111-1283-8743 (Other: World Health Organisation (WHO)); 2022-003384-24 (EudraCT Number); 2023-506825-13 (Other: EU CT Number)
Record Dates: First submitted 2023-05-29; First posted 2023-06-07 (Actual); Last update posted 2025-01-03 (Actual); Status verified 2025-01

CONDITIONS: Alzheimers Disease
MeSH Terms: conditions — Alzheimer Disease | interventions — semaglutide

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Study intervention period 1 (Experimental): Participants will receive either semaglutide or placebo matched to semaglutide once-weekly subcutaneous (s.c.) injections for 12 weeks as an add on therapy to standard of care. Participants initially received 0.25 milligram (mg) once weekly and the dose was then escalated once in 4 weeks until the maintenance dose (1.0 mg) was reached: 0.25 mg (week 1 to week 4), 0.5 mg (week 5 to week 8), 1.0 mg (week 9 to week 12).
  Interventions: Drug: Semaglutide; Drug: Placebo
- Study intervention period 2 (Placebo Comparator): All participants will receive 1.0 mg semaglutide s.c. injections once weekly for 52 weeks during study intervention period 2 as an add-on therapy to standard of care. Participants randomised to semaglutide s.c. 1.0 mg during study intervention period 1 remained on 1.0 mg target maintenance dose for 52 weeks from weeks 12-64. Participants initially randomised to placebo during study intervention period 1 will receive semaglutide s.c. in dose escalation fashion for 8 weeks (0.25 mg from weeks 12-16 and 0.5 mg from weeks 16-20) followed by a maintenance period from weeks 20-64 at dose 1.0 mg.
  Interventions: Drug: Semaglutide

INTERVENTIONS:
Drug: Semaglutide — Semagllutide will be administered once weekly subcutaneously.
Drug: Placebo — Placebo matched to semaglutide will be administered once weekly subcutaneously.
  Arms: Study intervention period 1

SUMMARY:
The study is being conducted to understand how the medicine, semaglutide, affects the immune system and other biological processes in people with Alzheimer's disease. Semaglutide is a medicine that doctors can prescribe in some countries for the treatment of type 2 diabetes and excess body weight. This study will help us understand whether semaglutide can also be used for the treatment of Alzheimer's disease. The study will last for about 77 weeks. In the first 12 weeks of treatment, participants will either get semaglutide (active medicine) or placebo (inactive dummy medicine). Which treatment participants get is decided by chance. In the following 52 weeks of treatment, all participants taking part in the study will get semaglutide. Participants must have a study partner, who is willing to take part in the study. Participants will get study medicine in a pen injector. The study partner will need to inject the study medicine into the skin of participant's stomach, thigh or upper arm once every week.

ELIGIBILITY:
Inclusion Criteria:

* Male or female, aged 55-75 years (both inclusive) at the time of signing the informed consent
* Mild cognitive impairment (MCI) or mild dementia of the Alzheimer's type according to the National Institute on Aging- Alzheimer's Association (NIA-AA) 2018 criteria
* Clinical dementia rating (CDR) global score of 0.5 or 1 at screening (visit 1)
* Amyloid positivity established with either historical amyloid positron emission tomography (PET) or historical cerebrospinal fluid (CSF) Aβ1-42 or historical CSF Aβ1-42/Aβ1-40 (historical data within the last 5 years) or blood sample for amyloid biomarker (Aβ42/Aβ40 ratio and p-tau217/np-tau217 ratio) at screening (visit 1)
* Treated with acetylcholinesterase inhibitors (approved for the treatment of Alzheimer's disease) and on stable dose for greater than 90 days before screening (visit 1)

Exclusion Criteria:

* Brain magnetic resonance imaging (MRI) scan suggestive of clinically significant structural central nervous system (CNS) disease confirmed by local read (example cerebral large-vessel disease [large vessel (cortical) infarcts greater than 10 millimeter (mm) in diameter], prior macro-haemorrhage [greater than 1centimeter cube (cm^3)], cerebral vascular malformations, cortical hemosiderosis, intracranial aneurism(s), intracranial tumours, changes suggestive of normal pressure hydrocephalus)
* Brain MRI scan suggestive of significant small vessel pathology confirmed by local read and defined as greater than 1 lacunar infarct and/or white matter hyperintensity (WMH) Fazekas13 scale greater than 2, (white matter [WM] greater than 20 mm) in the deep white matter and periventricular regions
* History or evidence of autoimmune diseases such as inflammatory bowel disease, rheumatoid arthritis, lupus, glomerulonephritis, psoriasis (but not limited to): Any other medical condition that would require use of systemic corticosteroids or immunosuppressants or immunostimulants in the 12 months prior to screening (visit 1)
* Received a vaccine product (including booster) 4 weeks prior to screening (visit 1) or expected to receive a vaccine product (including booster) before visit 5
* Use of any systemic immunomodulating drugs (small molecules and/or biologics) in the last 12 months prior to screening (visit 1) or anticipated use of such drugs during study intervention period 1 (i.e., during the first 12 weeks of treatment until visit 5), such as corticosteroids for systemic use, immunostimulants and immunosuppressants

Ages: 55 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 24 (Estimated)
Dates: Start 2023-06-20 (Actual); Primary Completion 2024-08-19 (Actual); Study Completion 2025-09-11 (Estimated)

PRIMARY OUTCOMES:
Change in gene expression assessed by single-cell ribonucleic acid sequencing (scRNAseq) (cells in cerebrospinal fluid [CSF]) | From baseline (week 0) to visit 5 (week 12)
  Measured as number of differentially expressed genes.
Change in gene expression assessed by scRNAseq (cells in blood) | From baseline (week 0) to visit 5 (week 12)
  Measured as number of differentially expressed genes.

SECONDARY OUTCOMES:
Number of treatment emergent adverse events (TEAEs) | From baseline (week 0) to visit 5 (week 12)
  Measured as count of events. An adverse event (AE) was defined as any unfavorable and unintended sign (including an abnormal laboratory finding), symptom or disease temporally associated with the use of a product, whether or not considered related to the product. A TEAE is defined as an event for which the onset of the event occurs during the treatment period.
Number of treatment emergent adverse events (TEAEs) | From baseline (week 0) to end of treatment (week 64)
  Measured as count of events. An adverse event (AE) was defined as any unfavorable and unintended sign (including an abnormal laboratory finding), symptom or disease temporally associated with the use of a product, whether or not considered related to the product. A TEAE is defined as an event for which the onset of the event occurs during the treatment period.
Weekly average semaglutide concentration (Cavg) based on population pharmacokinetic (PK) analysis | From visit 3 (week 4) to end of treatment (week 64)
  Measured in nanomoles per liter (nmol/L).

CONTACTS AND LOCATIONS:
Overall Officials: Clinical Transparency (dept. 2834), Study Director — Novo Nordisk A/S
Locations (10):
- United States (2):
  - Banner Sun Health Research Institute, Sun City, Arizona
  - Brain Matters Research, Delray Beach, Florida
- Canada (2):
  - Ottawa Memory Clinic, Ottawa, Ontario
  - Memory Program, Toronto, Ontario
- Rigshospitalet - afsnit 8015, København Ø, Denmark
- Italy (3):
  - Azienda Ospedaliera Spedali Civili di Brescia, Brescia
  - Azienda Ospedaliera di Perugia;Ospedale S. Maria della Miser, Perugia
  - Fondazione Santa Lucia IRCCS, Roma
- Karolinska Universitetssjukhuset, Huddinge, Stockholm, Sweden
- Centre de la Mémoire, Geneva, Switzerland

IPD SHARING:
Plan to Share IPD: Yes
According to the Novo Nordisk disclosure commitment on novonordisk-trials.com
URL: http://novonordisk-trials.com